CLINICAL TRIAL: NCT04282863
Title: Comparison Between Robotic (RM) and Laparoscopic Myomectomy (LM): a Multicenter Randomized Trial (RoLM Trial)
Brief Title: Comparison Between Robotic (RM) and Laparoscopic Myomectomy (LM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Tri-Service General Hospital (Other); Taipei Medical University WanFang Hospital (Other); Asian Society for Gynecologic Robotic Surgery (ASGRS) (Unknown)
Responsible Party: Principal Investigator, Hung-Cheng Lai, Vice President, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASGRS-TW001(RM:LM)
Record Dates: First submitted 2020-02-07; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Uterine Leiomyoma; Surgical Procedure, Unspecified
Keywords: Uterine Leiomyoma; robot-assisted (RM); conventional lapatoscopic myomectomy (LM)
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single-blinded RCT evaluating the effect of RM and LM in the management of uterine leiomyomas. Participants will be stratified on hospital performing the procedure and thereafter randomly assigned to the RM or LM group with allocation ratio 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic-assisted laparoscopic myomectomy (RM) (Active Comparator): After randomization, participants who are assigned to the robotic-assisted laparoscopic myomectomy (RM) agree to receive RM.
  Interventions: Procedure: RM
- Conventional laparoscopic myomectomy (LM) (Placebo Comparator): After randomization, participants who are assigned to the Conventional laparoscopic myomectomy (LM) agree to receive LM.
  Interventions: Procedure: LM

INTERVENTIONS:
Procedure: RM — All patients were positioned in a lithotomy position. A uterine manipulator and a Foley catheter were inserted. Four trocars were used after pneumoperitoneum was obtained. Trocar sites varied according to different procedures. Generally, umbilical site for the scope and 8-10 cm lateral to the scope at 15 degrees for the arms are the most commonly adopted sites for robotic myomectomy.
  Other Names: Robotic-assisted laparoscopic myomectomy
  Arms: robotic-assisted laparoscopic myomectomy (RM)
Procedure: LM — All patients were positioned in a lithotomy position. A uterine manipulator and a Foley catheter were inserted. Four trocars were used after pneumoperitoneum was obtained: a 10 mm port is inserted through the umbilicus to introduce the video-laparoscopic system. Other three accessory 5 mm trocar are inserted into the abdomen to the left lower quadrant, right lower quadrant, suprapubic area, for operative instruments and the suction irrigator cannula.
  Other Names: Conventional laparoscopic myomectomy
  Arms: Conventional laparoscopic myomectomy (LM)

SUMMARY:
This is a single-blinded RCT evaluating the effect of robotic-assisted (RM) or conventional laparoscopic surgery (LM) in the management of uterine leiomyomas.

DETAILED DESCRIPTION:
Uterine fibroids are the most common benign tumors of the uterus and may be presented 20%-40% of women at reproductive age.The uterine fibroids can be asymptomatic without intervention. However, they often are the cause of abnormal uterine bleeding, pelvic pain, infertility, and even miscarriage. Myomectomy, rather than hysterectomy can be one option for symptomatic women who wish to preserve their childbearing capabilities or for reasons other than for fertilit. Nowadays, patients pursue cosmetic benefit and early recovery and prompted the search for more conservative and minimally invasive surgical methods when surgical intervention is inescapable and surgical devices are improved.

The feasibility, safety and advantage of cosmetics of laparoscopic myomectomy (LM) has been confirmed after the improvement of techniques and instruments. However, it is very "unfriendly" for our surgeons because of many disadvantages such as keeping stand for long time, unable to relying on, or swaying visual field by first-assistant, etc. Since the approval by the US Food and Drug Administration (FDA) in April 2005, robotic surgeries using the da Vinci Surgical System (Intuitive surgical Inc., Sunnyvale, CA, USA) have been applied widely in many surgical fields including gynecology, urology, orthopedics, general surgery and cardiothoracic surgery. The three-dimensional vision system and the wrist-like structure of EndoWrist instruments (Intuitive surgical Inc., Sunnyvale, CA, USA) recapitulating the motion of the surgeon's hand make precise procedures easier than in conventional laparoscopy, which allows robotic surgery to overcome some of the shortcomings and limitations of traditional laparoscopy. Dr. Lai and colleagues had also successfully undergone robotic surgery in many complicated gynecologic diseases in Taiwan.

However, how to choose or apply robotic-assisted (RM) or conventional laparoscopic surgery (LM) in the management of uterine leiomyomas is still an important issue for our surgeon. We still lack clear definitions about which one kind of myoma may be smoothly performed in RM or LM. The current study is aimed to compare the clinical outcome and efficacy of these 2 minimally invasive procedure in myomectomy, RM and LM, for women with symptomatic uterine fibroids, in this prospective randomised control trial.

ELIGIBILITY:
Inclusion Criteria:

* All women who has symptomatic benign myoma.

Exclusion Criteria:

* Patient is unwilling the scheduled operation after randomization.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The women, age more than 20 y/o, have symptomatic benign myoma.
Enrollment: 494 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | The surgical 1 day
  To compare the conversion rate between RM and LM

SECONDARY OUTCOMES:
The time of surgery | The surgical 1 day
The amount of blood loss and transfusion | Through hospitalization duration, an average of 1 week
The dosage of antipyretic | Through hospitalization duration, an average of 1 week
The stay length of hospitalization | Through hospitalization duration, an average of 1 week
Readmission rate | Within 1 month after discharge
Myoma score | Through study completion, an average of 2 years
  The score of myoma characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chang Lai, M.D/Ph. D., Principal Investigator — Study Principal Investigator
Locations (1):
- Taipei Medical University Shuang Ho Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No